CLINICAL TRIAL: NCT00190294
Title: Comparison Expectant With Immediate Medical Management for the Evacuation of the no Evolutionary Pregnancies Before 13 GW
Brief Title: Expectant Versus Immediate Medical Management for the Evacuation of the no Evolutionary Pregnancies Before 13 GW
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Isabelle Brindel, Department Clinical Research of developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P011017
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2007-03

CONDITIONS: Pregnancy Complications
Keywords: Pregnancy Complications
MeSH Terms: conditions — Pregnancy Complications | interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): MIFEPRISTONE 200 mg and misoprostol 400 µg
  Interventions: Drug: MIFEPRISTONE 200 mg and misoprostol 400 µg

INTERVENTIONS:
Drug: MIFEPRISTONE 200 mg and misoprostol 400 µg — MIFEPRISTONE 200 mg and misoprostol 400 µg

SUMMARY:
Compared the interest of one week expectancy vs immediate medical treatment in the taking care of the evacuation of the no evolutionary pregnancies before 13 GW.

DETAILED DESCRIPTION:
Randomized control trial comparing one week expectancy vs immediate medical treatment (mifepristone 200mg and misoprostol 400ug) in the taking care of the evacuation of the no evolutionary pregnancies before 13 GW.

ELIGIBILITY:
Inclusion Criteria:

* Agreed women aged over 18 yrs old

Non evolutive pregnancy before 13GW :

* Non evolutive pregnancy with no fetal cardiac activity
* Non evolutive pregnancy with embryonic structures
* Trophoblastic material in uterine cavity P bhCG < 10UI/L

Exclusion criteria:

* Age < 18 years
* pregnancy evolutionary
* not evolutionary pregnancy after 13 weeks of amenorrhoea characterized by the presence of an scan image intra-uterine ANECHOGENE furthermore of 50mm of diameter
* amenorrhoea of more than 13 weeks
* pregnancy twin
* pregnancy molar
* pregnancy extra-uterine
* Extra-uterine pregnancy
* one or many contraindications in the mifepristone:
* Allergy known about the MIFEPRISTONE
* Incapacity suprarenal
* corticosteroid therapy in the long price
* confusions of the haemostasis (thrombopenia < in 100000 / mm3)
* anaemia (rate Hg < in 9 g / dl)
* contraindication in the misoprostol
* allergy known about PROSTAGLANDINES
* BEANCE cervical

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2003-04; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Number of surgical evacuation in each group | during de study
  Number of surgical evacuation in each group

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Rosenberg, Study Chair — Poissy Hospital
Locations (1):
- Poissy Hospital, Poissy, France

REFERENCES:
- [Derived] Ghosh J, Papadopoulou A, Devall AJ, Jeffery HC, Beeson LE, Do V, Price MJ, Tobias A, Tuncalp O, Lavelanet A, Gulmezoglu AM, Coomarasamy A, Gallos ID. Methods for managing miscarriage: a network meta-analysis. Cochrane Database Syst Rev. 2021 Jun 1;6(6):CD012602. doi: 10.1002/14651858.CD012602.pub2. PMID 34061352
- [Derived] Torre A, Huchon C, Bussieres L, Machevin E, Camus E, Fauconnier A. Immediate versus delayed medical treatment for first-trimester miscarriage: a randomized trial. Am J Obstet Gynecol. 2012 Mar;206(3):215.e1-6. doi: 10.1016/j.ajog.2011.12.009. Epub 2011 Dec 16. PMID 22381604